CLINICAL TRIAL: NCT02919007
Title: Clinical Evaluation of Silk'n HST Self-selection, Labeling Comprehension, and Device Use
Brief Title: Silk'n HST Device Usability and Self Selection Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO111411
Record Dates: First submitted 2016-09-25; First posted 2016-09-29 (Estimated); Results first posted 2018-09-27 (Actual); Last update posted 2018-10-31 (Actual); Status verified 2016-09

CONDITIONS: Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silk'n HST treatment (Experimental): Intervention includes treatment with the Silk'n HST on the periorbital areas as instructed in the user's manual. Measure includes the ability to operate the device correctly according to the user manual.
  Interventions: Device: Silk'n HST treatment

INTERVENTIONS:
Device: Silk'n HST treatment — Intervention includes treatment with the Silk'n HST on the periorbital areas as instructed in the user's manual

SUMMARY:
This is a Usability study, conducted for the purpose of testing Silk'n HST Device usability.

DETAILED DESCRIPTION:
Study objectives:

To test the Silk'n HST Device usability, i.e., the self-selection, labeling comprehension, and safe and effective device use by potential end users, under actual use conditions. Additionally, this study was aimed to evaluate if contraindicated subjects self-exclude from use of the device.

Investigation Design:

The study is a usability study. Twenty five potential participants were enrolled in a single location (shopping mall). Participants received the Silk'n HST device in its original package with the complete user manual and performed a full treatment. Post-treatment questionnaire and labeling comprehension exam were conducted following treatment. Out of the twenty five subjects five participants contraindicated to the study inclusion criteria were self-exclude from use of the device.

Success criteria:

Using the device, all 20 tested subjects are able to complete device related tasks, including applying and operating the Silk'n device without assistance in a timeframe of up to one hour and with minimal attempts to ask for assistance.

Additionally, measurable usability criteria for specific, critical steps, such as time-to-completion, frequency of attempts to ask examiner, numerical ratings, etc., were evaluated using observer evaluation and user post-test questionnaire responses.

Sample Size:

Twenty five subjects identified as potential end users of the device including five subjects with contraindication to the device were recruited to the study. The number of subjects is appropriate considering the device and user related risks, low probable occurrence and severity of these risks, and the design of the study. Furthermore, usability studies are not seeking statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female equal to or greater than 18 years of age.
* Subject is a potential candidate for purchasing the Silk'n HST device.
* Subject has facility with both hands.
* Subject is capable of understanding and is willing to sign informed consent.

Exclusion Criteria:

* Subject with dark brown or black spots, such as large freckles, birth marks, moles or warts on the area to be treated.
* Subject with eczema, psoriasis, lesions, open wounds or active infections, such as cold sore in the area to be treated.
* Subject with a history of kelodial scar formation, a known sensitivity to light (photosensitivity) or is taking medication that makes the skin more sensitive to light, including non-steroidal anti-inflammatory agents, (e.g., aspirins, ibuprofens, acetaminophen), tetracyclines, phenothiazines, thiazide, diuretics, sulfonyluraes, sulfonamides, DTIC, fluorouracil, vinblastine, griseofulvin, Alpha-Hydroxi Acids (AHAs), Beta-Hydroxi Acids (BHAs), Retin-A®, Accutane® and/or topical retinoids.
* Subject with abnormal skin conditions caused by diabetes, for example, or other systemic or metabolic diseases.
* Subject currently or has recently been treated with Alpha-Hydroxi Acids (AHAs), Beta-Hydroxi Acids (BHAs), Retin-A®, topical retinoids or azelaic acid.
* Subject has been treated with Accutane® (isotretinoin) within the past 6 months.
* Subject has been on a steroid regimen within the past 3 months.
* Subject has a history of herpes outbreaks in the area of treatment.
* Subject suffers from epilepsy.
* Subject with an active implant, such as a pacemaker, incontinence device, insulin pump, etc.
* Subject with a disease related to photosensitivity, such as porphyria, polymorphic light eruption, solar urticaria, lupus, etc.
* Subject with a history of skin cancer or areas of potential skin malignancies.
* Subject received radiation therapy or chemotherapy treatments within the past 3 months.
* Subject is pregnant or nursing (lactating).

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Silk'h HST Treatment: Intervention includes treatment with the Silk'n HST on the periorbital areas as instructed in the user's manual. Measure includes the ability to operate the device correctly according to the user manual.
  Silk'h HST treatment: Intervention includes treatment with the Silk'n HST on the periorbital areas as instructed in the user's manual
Period: Overall Study
Arm/Group | Silk'h HST Treatment
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Silk'h HST Treatment
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (15.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Usability Assessment
Description: Study success is determined according to the ability of all subjects to complete device related tasks, including applying and operating the Device without assistance in a timeframe of up to 1 hour and with minimal attempts to ask for assistance.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Arm/Group | Silk'n HST Treatment
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Arm/Group | Silk'h HST Treatment
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No